CLINICAL TRIAL: NCT02227654
Title: Evaluating the Performance of Morphology Index in Surgical Decision-Making for Ovarian Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederick R. Ueland, M.D. (Other)
Collaborators: Lucille P. Markey Cancer Center at University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Frederick R. Ueland, M.D., Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-GYN-200
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Ovarian Neoplasms
Keywords: Ovary; Cancer; Morphology; Surgery
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abnormal Ovarian Ultrasound (Experimental): Abnormal Ovarian Ultrasound
  Interventions: Procedure: Abnormal Ovarian Ultrasound

INTERVENTIONS:
Procedure: Abnormal Ovarian Ultrasound — Ultrasound

SUMMARY:
The present investigation will prospectively evaluate whether serial transvaginal ultrasonography with Morphology Index (MI) can further reduce false positive results by more accurately distinguishing benign from malignant ovarian tumors. If there is no change in the detection of true positive cases, the result will be an increase in the positive predictive value of ovarian cancer screening.

DETAILED DESCRIPTION:
Primary Objective:

To determine if a treatment algorithm using serial transvaginal ultrasound with a tumor morphology index can improve the positive predictive value (PPV) of ovarian cancer screening compared to a historical control from 15% to 25%.

Secondary Objective To measure the compliance for study participants enrolled on the treatment algorithm using serial transvaginal ultrasound with a tumor morphology index.

Exploratory Objective To determine the effectiveness of a treatment algorithm that combines serum biomarkers aloneor in combination with transvaginal ultrasound to reduce the false positive rate of ovarian cancer screening in the subset of women agreeing to biomarker collection.

ELIGIBILITY:
Inclusion Criteria:

* Women must be enrolled in the University of Kentucky Ovarian Cancer Screening Program Eligibility criteria for the OCSP are: 50 years of age or older, or be postmenopausal and have not had a prior salpingo-oophorectomy or have a family history of ovarian cancer in a primary relative or have a self-history of breast cancer.
* Patients have a documented ovarian abnormality on ultrasound
* Patients having undergone prior hysterectomy will be eligible provided that they meet the other requirements for entry into this study.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who are not enrolled in the University of Kentucky Ovarian Cancer Screening Program .
* Patients who cannot tolerate the vaginal ultrasound procedure.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who are referred with pelvic symptoms, a known pelvic mass, or a history of prior radiation, will be excluded from this investigation.
* History of ovarian cancer.
* Prior bilateral salpingo-oophorectomy.
* Prisoners.
* Women who are currently pregnant.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Because ovarian cancer is a disease of only women, men are not included in this study, but women of all races and ethnic groups are eligible for this trial.
Enrollment: 179 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Positive predictive value (PPV) of ovarian cancer screening | Up to 12 months
  Whether the treatment algorithm for patients with abnormal ultrasounds improves the positive predictive value of ultrasounds as ovarian screening tests, thus lowering the false positive rate compared to historical controls.

SECONDARY OUTCOMES:
Surgical complications | Up to 12 months
  Surgical complications including type, severity, and resolution.
Compliance to the treatment algorithm | Up to 12 months
  Percentage of required visits that were attended for each individual's treatment algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R. Ueland, M.D., Principal Investigator — Markey Cancer Center, University of Kentucky
Locations (1):
- Markey Cancer Center, University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No